CLINICAL TRIAL: NCT03479879
Title: Estradiol Pretreatment With Misoprostol in Second Trimester Miscarriage: A Prospective, Double-blind, Randomized Clinical Trial
Brief Title: Estradiol Pretreatment With Misoprostol in Second Trimester Miscarriage
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS1731
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Estradiol; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Estradiol + Misoprostol (Experimental)
  Interventions: Drug: Estradiol; Drug: Misoprostol
- Placebo + Misoprostol (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet; Drug: Misoprostol

INTERVENTIONS:
Drug: Estradiol — Estradiol
  Arms: Estradiol + Misoprostol
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo + Misoprostol
Drug: Misoprostol — Misoprostol

SUMMARY:
To compare the effectiveness of estradiol pretreatment with misoprostol and vaginal misoprostol alone in induction of second trimestr miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age more than 18 years old (age of legal consent).
* Gestational age between 12-26 weeks.
* Hb level > 10 g/dL.
* BMI between 25 kg/m2 and 35 kg/m2.
* Missed abortion.
* Living fetus with multiple congenital malformations incompatible with life.
* PPROMS with drained liquor and parents are consenting for termination of pregnancy.

Exclusion Criteria:

* Maternal age less than 18 years old.
* Gestational age less than 12 weeks or more than 26 weeks.
* Hb level < 10 g/dL.
* Scared uterus (previous myomectomy - cesarean section - hysterectomy and ruptured uterus).
* Polyhydramnios.
* Anencephaly.
* Fibroid uterus.
* BMI less than 25 kg/m2 and more than 35 kg/m2.
* Coagulopathy.
* Previous attempts for induction of abortion in the current pregnancy.
* Allergy to misoprostol or estradiol.
* Placenta previa.
* Medical disorder that contraindicate induction of abortion (e.g. heart failure).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Duration of induction of abortion | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt